CLINICAL TRIAL: NCT05136950
Title: Incidence of Glaucoma-related Adverse Events in Pediatric Secondary Intraocular Lens Implantation, In-the-bag Versus Sulcus Fixation : a Randomized Controlled Trial
Brief Title: Incidence of Glaucoma-related Adverse Events in Pediatric Secondary Intraocular Lens Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021KYPJ135
Record Dates: First submitted 2021-11-01; First posted 2021-11-30 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Lens Implantation, Intraocular
Keywords: Pediatric aphakia; Secondary Intraocular Lens Implantation; Glaucoma-related Adverse Events; In-the-bag IOL implantation; Sulcus IOL fixation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secondary in-the-bag IOL fixation group (Experimental): In-the-bag IOL fixation is the experimental arm
  Interventions: Procedure: Secondary in-the-bag IOL fixation
- Secondary ciliary sulcus IOL fixation group (Active Comparator): Ciliary sulcus IOL fixation is the control arm
  Interventions: Procedure: Secondary ciliary sulcus IOL fixation

INTERVENTIONS:
Procedure: Secondary in-the-bag IOL fixation — The experimental group with secondary IOL fixated in the capsular bag
  Arms: Secondary in-the-bag IOL fixation group
Procedure: Secondary ciliary sulcus IOL fixation — The control group with secondary IOL fixated in the ciliary sulcus
  Arms: Secondary ciliary sulcus IOL fixation group

SUMMARY:
To compare the incidence of glaucoma-related adverse events of in-the-bag versus ciliary-sulcus-fixed secondary intraocular lens (IOL) implantation in pediatric aphakia

DETAILED DESCRIPTION:
Treatment of pediatric cataract, one of the leading causes of childhood blindness globally, remains challenging because of extremely high incidence of glaucoma-related adverse events (AEs) after IOL implantation. The investigators aim to compare the incidence of glaucoma-related AEs of in-the-bag versus ciliary-sulcus-fixed secondary intraocular lens (IOL) implantation in pediatric aphakia.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 months and 14 years
* Had a primary diagnosis of congenital cataract.
* Underwent cataract extraction between the ages of 2 and 24 months

Exclusion Criteria:

* Primary IOL implantation
* Pre-existing ocular disease which might affect the location and outcome of secondary IOL implantation (including and not restricted to microphthalmia, microcornea, microcornea, corneal opacity, pseudopterygium, iris anomaly, glaucoma diagnosed before cataract extraction, uveitis, persistent fetal vasculature or trauma)
* Suture fixation for secondary IOL implantation

Ages: 18 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2033-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of glaucoma-related adverse events | One year after surgery
  The assessment of glaucoma-related adverse events is performed at one year after surgery

SECONDARY OUTCOMES:
Incidence of glaucoma-related adverse events | Six months,three years, five years, ten years after surgery
  The assessment of glaucoma-related AEs is performed at six months, three years, five years, ten years after surgery
Visual acuity | Six months,one year, three years, five years, ten years after surgery
  Evaluated with an ETDRS chart. For those who are unable to use ETDRS chart, visual acuity will be evaluated with Lea Symbol Chart or Teller Acuity Cards
Ocular refractive power | Six months,one year,three years, five years, ten years after surgery
  Measured by the Auto Refractometer
Intraocular lens decentration | Six months,one year, three years, five years, ten years after surgery
  Measured by anterior segment scanning
Intraocular lens tilt | Six months,one year, three years, five years, ten years after surgery
  Measured by anterior segment scanning
Incidence of other adverse events | Six months,one year, three years, five years, ten years after surgery
  The assessment of other adverse events will be performed at six months,one year,three years, five years, ten years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, PhD, Principal Investigator — Zhongshan Ophthalmic center, Guangzhou, People's Republic of China
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University Guangzhou, China, 510060, Guangzhou, China

REFERENCES:
- [Result] Liu Z, Lin H, Jin G, Tan X, Qu B, Jin L, Chen X, Wang W, Han X, Xu J, Ying G, Han Y, He M, Congdon N, Chen W, Luo L, Liu Y. In-the-Bag Versus Ciliary Sulcus Secondary Intraocular Lens Implantation for Pediatric Aphakia: A Prospective Comparative Study. Am J Ophthalmol. 2022 Apr;236:183-192. doi: 10.1016/j.ajo.2021.10.006. Epub 2021 Oct 13. PMID 34653355
- [Result] Wood KS, Tadros D, Trivedi RH, Wilson ME. Secondary intraocular lens implantation following infantile cataract surgery: intraoperative indications, postoperative outcomes. Eye (Lond). 2016 Sep;30(9):1182-6. doi: 10.1038/eye.2016.131. Epub 2016 Jul 1. PMID 27367747
- [Result] Freedman SF, Beck AD, Nizam A, Vanderveen DK, Plager DA, Morrison DG, Drews-Botsch CD, Lambert SR; Infant Aphakia Treatment Study Group. Glaucoma-Related Adverse Events at 10 Years in the Infant Aphakia Treatment Study: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2021 Feb 1;139(2):165-173. doi: 10.1001/jamaophthalmol.2020.5664. PMID 33331850
- [Result] Shenoy BH, Mittal V, Gupta A, Sachdeva V, Kekunnaya R. Complications and visual outcomes after secondary intraocular lens implantation in children. Am J Ophthalmol. 2015 Apr;159(4):720-6. doi: 10.1016/j.ajo.2015.01.002. Epub 2015 Jan 9. PMID 25579641
- [Result] Zhao YE, Gong XH, Zhu XN, Li HM, Tu MJ, Coursey TG, Pflugfelder SC, Gu F, Chen D. Long-term outcomes of ciliary sulcus versus capsular bag fixation of intraocular lenses in children: An ultrasound biomicroscopy study. PLoS One. 2017 Mar 16;12(3):e0172979. doi: 10.1371/journal.pone.0172979. eCollection 2017. PMID 28301497
- [Result] Whitman MC, Vanderveen DK. Complications of pediatric cataract surgery. Semin Ophthalmol. 2014 Sep-Nov;29(5-6):414-20. doi: 10.3109/08820538.2014.959192. PMID 25325868
- [Derived] Zou Y, Jin L, Qu B, Chen H, Zeng M, Li X, Liu X, Luo L, Liu Z, Liu Y. Safety and efficacy in pediatric secondary intraocular lens implantation, in-the-bag versus sulcus implantation: a multicenter, single-blinded randomized controlled trial. Trials. 2023 Jun 9;24(1):388. doi: 10.1186/s13063-023-07411-z. PMID 37296411